CLINICAL TRIAL: NCT00891046
Title: An Open-label Extension Study of Canakinumab (ACZ885) in Patients With Systemic Juvenile Idiopathic Arthritis (SJIA) and Active Systemic Manifestations Who Participated in Studies ACZ885G2301 and ACZ885G2305; and Response Characterization Study in Canakinumab Treatment-naïve Patients With Active SJIA With and Without Fever
Brief Title: An Open-label Extension Study of Canakinumab in Patients With Systemic Juvenile Idiopathic Arthritis and Active Systemic Manifestations Manifestations and Response Characterization Study in Canakinumab Treatment-naïve Patients With Active SJIA With and Without Fever.
Acronym: β-SPECIFIC 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Pediatric Rheumatology International Trials Organization (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885G2301E1; EudraCT: 2008-008008-42
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2018-07

CONDITIONS: Systemic Juvenile Idiopathic Arthritis
Keywords: Flare; arthritis; IL-1beta antagonist; systemic juvenile idiopathic arthritis; CHAQ; steroids; ACR pediatric response; Systemic juvenile idiopathic arthritis with active flare
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — canakinumab

ARMS (1):
- Canakinumab (Experimental): Canakinumab
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab — Canakinumab

SUMMARY:
This open-label extension study will permit patients with Systemic Juvenile Idiopathic Arthritis (SJIA) who previously were responsive to treatment with canakinumab and canakinumab treatment-naïve patients with active SJIA with and without fever to be retreated with 4 mg/kg s.c. every 4 weeks and assessed for continued efficacy and safety until discontinuation or when study CACZ885G2402 is in place at their study center or around March 2013, whichever occurs first. Patients who are steroid-free will be able to taper their canakinumab dose to 2 mg/kg s.c. every 4 weeks.

ELIGIBILITY:
Inclusion criteria:

* Patients from study CACZ885G2305 or CACZ885G2301 who achieved an adapted ACR pediatric 30 response 15 days after their initial dose of canakinumab but clinically deteriorated afterwards or a minimum ACR Pediatric 30 response was not maintained after Day 15 and intervention is deemed necessary by the investigator, or Patients in study CACZ885G2301 who are not eligible to enter Part II (withdrawal part) because they were not able to meet the corticosteroid entry criteria , or Responder patients in Part I or Part II who had not flared when CACZ885G2301 was stopped, or CACZ885G2301 patients who were responders in Part I but experienced a flare in Part II.
* Treatment-naïve patients need to meet the following criteria:

  * Confirmed diagnosis of systemic juvenile idiopathic arthritis as per ILAR definition that must have occurred at least 2 months prior to enrollment with onset of disease < 16 years of age
  * Male and female patients aged ≥ 2 to < 20 years of age
  * Active disease at the time of enrollment defined as having 2 or more of the following:

    * Documented spiking, intermittent fever (body temperature > 38°C) for at least 1 day during the screening period and within 1 week before first canakinumab dose
    * At least 2 joints with active arthritis
    * AND C-reactive protein (CRP) > 30 mg/L (normal range < 10 mg/L) Rash Serositis Lymphadenopathy Hepatosplenomegaly
  * Naïve to canakinumab

Other protocol-defined inclusion criteria may apply

Exclusion criteria:

* History of allergy or hypersensitivity to study drug
* With active or recurrent bacterial, fungal or viral infections at time of enrollment

Other protocol inclusion/exclusion criteria may apply

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 270 (Actual)
Dates: Start 2009-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (67):
- United States (6):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Portland, Oregon
- Novartis Investigative Site, CABA, Buenos Aires, Argentina
- Novartis Investigative Site, Vienna, Austria
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Laken
  - Novartis Investigative Site, Leuven
- Brazil (3):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (4):
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Strasbourg
- Germany (11):
  - Novartis Investigative Site, Bad Bramstedt
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Garmisch-Partenkirchen
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Saint Augustin
  - Novartis Investigative Site, Tübingen
- Greece (3):
  - Novartis Investigative Site, Ampelokipoi, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Goudi- Athens
- Novartis Investigative Site, Budapest, Hungary
- Israel (5):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
- Italy (4):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Utrecht, Netherlands
- Novartis Investigative Site, Breña, Lima region, Peru
- Novartis Investigative Site, Warsaw, Poland
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (3):
  - Novartis Investigative Site, Esplugues de Llobregat, Barcelona
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Lausanne, Switzerland
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Balcova / Izmir
  - Novartis Investigative Site, Fatih / Istanbul
  - Novartis Investigative Site, Istanbul
- United Kingdom (7):
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Newcastle Upon Tyme
  - Novartis Investigative Site, Oxford

REFERENCES:
- [Derived] Ruperto N, Brunner HI, Quartier P, Constantin T, Wulffraat NM, Horneff G, Kasapcopur O, Schneider R, Anton J, Barash J, Berner R, Corona F, Cuttica R, Fouillet-Desjonqueres M, Fischbach M, Foster HE, Foell D, Radominski SC, Ramanan AV, Trauzeddel R, Unsal E, Levy J, Vritzali E, Martini A, Lovell DJ; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Canakinumab in patients with systemic juvenile idiopathic arthritis and active systemic features: results from the 5-year long-term extension of the phase III pivotal trials. Ann Rheum Dis. 2018 Dec;77(12):1710-1719. doi: 10.1136/annrheumdis-2018-213150. Epub 2018 Sep 29. PMID 30269054
- [Derived] Grom AA, Ilowite NT, Pascual V, Brunner HI, Martini A, Lovell D, Ruperto N; Paediatric Rheumatology International Trials Organisation and the Pediatric Rheumatology Collaborative Study Group; Leon K, Lheritier K, Abrams K. Rate and Clinical Presentation of Macrophage Activation Syndrome in Patients With Systemic Juvenile Idiopathic Arthritis Treated With Canakinumab. Arthritis Rheumatol. 2016 Jan;68(1):218-28. doi: 10.1002/art.39407. PMID 26314396
- See also: Related Info — http://www.novartisclinicaltrials.com
- See also: Related Info — http://www.juvenilearthritisresearch.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 61 centres in 20 countries.
Pre-assignment Details: A total of 147 participants from studies CACZ885G2301 (NCT number: NCT00889863) and CACZ885G2305 (NCT number: NCT00886769) and 123 canakinumab treatment- naive participants were enrolled into this extension study.
Groups:
- ACZ885 Treated: Group 1 (Discontinued From Core Study): Participants who discontinued from Study CACZ885G2301 Part 2 (NCT00889863) due to SJIA flare, received a subcutaneous (s.c.).
- ACZ885 Treated: Group 2 (Completed Core Study): Participants who completed Study CACZ885G2301 (NCT00889863), received an s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study): Participants who failed to taper their steroid dose in CACZ885G2301 (NCT00889863); received an s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treated: Group 4 (Other Criteria): Participants who previously received canakinumab treatment in Studies CACZ885G2301 (NCT00889863) and CACZ885G2305 (NCT00886769), but did not fulfill the criteria for Group 1, 2 or 3, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treatment Naive: Participants who were canakinumab treatment naive and did not participate in previous canakinumab studies, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
Period: Overall Study
Arm/Group | ACZ885 Treated: Group 1 (Discontinued From Core Study) | ACZ885 Treated: Group 2 (Completed Core Study) | ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study) | ACZ885 Treated: Group 4 (Other Criteria) | ACZ885 Treatment Naive
Started | 33 | 63 | 40 | 11 | 123
Completed | 21 | 54 | 17 | 8 | 84
Not Completed | 12 | 9 | 23 | 3 | 39
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 5 | 2 | 19 | 2 | 20
Not completed — Administrative problems | 0 | 0 | 0 | 0 | 1
Not completed — Participant no longer required drug | 0 | 2 | 0 | 0 | 1
Not completed — Adverse Event | 4 | 3 | 2 | 0 | 14
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set: The analysis was performed in safety set (SAF), defined as all participants who received at least one dose of study drug.
Groups:
- ACZ885 Treated: Group 1 (Discontinued From Core Study): Participants who discontinued from NCT00889863, received a subcutaneous (s.c.) injection of canakinumab 4 mg/kg every 4 weeks unless discontinuation occurs. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treated: Group 2 (Completed Core Study): Participants who completed study NCT00889863, received an s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study): Participants who failed to taper their steroid dose in NCT00889863; received an s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treated: Group 4 (Other Criteria): Participants who previously received canakinumab treatment in Studies NCT00889863 and NCT00886769, but did not fulfill the criteria for Group 1, 2 or 3, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treatment Naive: Participants who were canakinumab treatment- naive and did not participate in previous canakinumab studies, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- Total: Total of all reporting groups
Arm/Group | ACZ885 Treated: Group 1 (Discontinued From Core Study) | ACZ885 Treated: Group 2 (Completed Core Study) | ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study) | ACZ885 Treated: Group 4 (Other Criteria) | ACZ885 Treatment Naive | Total
Number analyzed (Participants) | 33 | 63 | 40 | 11 | 123 | 270
Age, Customized [Number; unit: participants]
  2 -- <4 years | 0 | 2 | 3 | 1 | 18 | 24
  4 -- <6 years | 6 | 10 | 6 | 5 | 15 | 42
  6 -- <12 years | 16 | 32 | 21 | 3 | 50 | 122
  12 -- <20 years | 11 | 17 | 10 | 2 | 40 | 80
  ≥ 20 years | 0 | 2 | 0 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 34 | 23 | 5 | 75 | 156
  Male | 14 | 29 | 17 | 6 | 48 | 114

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), AEs by Severity, AEs Leading to Discontinuation, SAEs Leading to Discontinuation, Treatment Related AEs and SAE
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not related to study drug. A SAE was defined as an event which was fatal or life threatening, required or prolonged hospitalization, was significantly or permanently disabling or incapacitating, constituted a congenital anomaly or a birth defect, or encompassed any other clinically significant event that could jeopardize the participants or require medical or surgical intervention to prevent one of the aforementioned outcomes. Treatment related AEs or SAEs were defined as AEs or SAEs that were suspected to be related to study treatment as per investigator.
Time Frame: From start of study treatment (Day 1) up to end of follow-up period (Week 271 for ACZ885 treated participants and Week 145 for ACZ885 treatment naive participants)
Population: The analysis was performed in safety set (SS), defined as all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- ACZ885 Treated: Participants who were responsive to canakinumab in previous studies: NCT00889863 and NCT00886769 and entered into this extension study in Group 1, 2, 3 and 4.
Arm/Group | ACZ885 Treatment Naive | ACZ885 Treated
Number analyzed (Participants) | 123 | 147
participants
  AEs | 108 | 137
  SAEs | 40 | 47
  Discontinuation due to any AE | 14 | 18
  Discontinuation due to any SAE | 13 | 14
  Treatment Related AEs | 44 | 57
  Treatment related SAEs | 1 | 4

2. Primary Outcome: Number of Participants With Anti -ACZ885 Antibodies at Any Visit During the Study
Description: Immunogenicity assessment included determination of anti-canakinumab (ACZ885) antibodies in serum samples using BIAcore system.
Time Frame: as for outcome 1
Population: The analysis was performed on the SS population.
Measure: Number; unit: participants
Arm/Group | ACZ885 Treatment Naive | ACZ885 Treated
Number analyzed (Participants) | 123 | 147
participants | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Local Injection Site Reactions During the Study
Description: Local injection site tolerability was assessed on the injection site. Each participant was classified into one of the following four categories: 1. no tolerability reactions at any time during the study, 2. mild reaction observed on at least one occasion but no moderate or severe reactions. 3. moderate reaction observed on at least one occasion but no severe reaction. 4. severe reaction observed on at least one occasion.
Time Frame: as for outcome 1
Population: The analysis was performed in SS population.
Measure: Number; unit: participants
Arm/Group | ACZ885 Treatment Naive | ACZ885 Treated
Number analyzed (Participants) | 123 | 147
participants
  No tolerability reaction | 115 | 129
  Mild tolerability reaction | 6 | 15
  Moderate tolerability reaction | 2 | 3
  Severe tolerability reaction | 0 | 0

4. Primary Outcome: Percentage of Participants Previously Treated With Anakinra Who Achieved Minimum Response of American College of Rheumatology (ACR) Pediatric 30/50/70/90/100 at Last Assessment of Study
Description: Adapted ACR Paediatric 30/50/70/90 or 100 was assessed based on following 7 variables: 1.Physician's Global Assessment on a 1-100 millimeter (mm) visual analog scale (VAS); 2. Participants Global Assessment on a 1-100 mm VAS; 3. Functional ability; 4. Joints count with active arthritis; 5. Joints count with limitation of motion; 6. Laboratory measure of C-reactive protein (CRP) and 7. Absence of intermittent fever due to severe juvenile idiopathic arthritis (SJIA) during the preceding week. Response was defined as more than or equal to (≥) 30%/50%/70%/90% or 100% improvement in at least 3 of the response variables 1 to 6, no intermittent fever (i.e. body temperature less than or equal to (≤) 38 °C) in the preceding week (variable 7) and with no more than one variable 1 to 6, worsening by more than 30%.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was done in FAS population. Here 'Number of participants analyzed' signifies number of participants with an ACR assessment at the given visit.
Measure: Number; unit: Percentage of participants
Groups:
- ACZ885 Treatment Naive: Group 1: Participants who were canakinumab treatment naive and who discontinued anakinra due to lack of efficacy, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treatment Naive: Group 2; ACZ885 Treatment Naive: Group 3: Participants who were canakinumab treatment naive and who discontinued anakinra for safety/tolerability reasons, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treatment Naive: Group 4: Participants who were canakinumab treatment naive and who never exposed to anakinra, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
Arm/Group | ACZ885 Treatment Naive: Group 1 | ACZ885 Treatment Naive: Group 2 | ACZ885 Treatment Naive: Group 3 | ACZ885 Treatment Naive: Group 4
Number analyzed (Participants) | 26 | 12 | 13 | 70
Percentage of participants
  ACR ≥30 criteria | 80.8 | 91.7 | 100 | 95.7
  ACR ≥ 50 criteria | 80.8 | 91.7 | 100 | 92.9
  ACR ≥ 70 criteria | 76.9 | 91.7 | 92.3 | 90
  ACR ≥ 90 criteria | 69.2 | 91.7 | 76.9 | 80
  ACR 100 criteria | 57.7 | 91.7 | 69.2 | 64.3

5. Primary Outcome: Percentage of Participants Previously Treated With Tocilizumab Who Achieved Minimum Response of American College of Rheumatology (ACR) Pediatric 30/50/70/90/100 at Last Assessment of Study
Description: Adapted ACR Paediatric 30/50/70/90 or 100 was assessed based on following 7 variables: 1.Physician's Global Assessment on a 0-100 mm VAS; 2. Participants Global Assessment on a 0-100 mm VAS; 3. Functional ability; 4. Joints count with active arthritis; 5. Joints count with limitation of motion; 6. Laboratory measure of CRP and 7. Absence of intermittent fever due to SJIA during the preceding week. Response was defined as ≥ 30%/50%/70%/90% or 100% improvement in at least 3 of the response variables 1 to 6, no intermittent fever (i.e. body temperature ≤ 38 °C) in the preceding week (variable 7) and with no more than one variable 1 to 6, worsening by more than 30%.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Groups:
- ACZ885 Treatment Naive: Group 1: Participants who were canakinumab treatment naive and who discontinued tocilizumab due to lack of efficacy, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treatment Naive: Group 2; ACZ885 Treatment Naive: Group 3: Participants who were canakinumab treatment naive and who discontinued tocilizumab for safety/tolerability reasons, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treatment Naive: Group 4: Participants who were canakinumab treatment naive and who never exposed to tocilizumab, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
Arm/Group | ACZ885 Treatment Naive: Group 1 | ACZ885 Treatment Naive: Group 2 | ACZ885 Treatment Naive: Group 3 | ACZ885 Treatment Naive: Group 4
Number analyzed (Participants) | 26 | 3 | 2 | 90
Percentage of participants
  ACR ≥30 criteria | 92.3 | 100 | 100 | 92.2
  ACR ≥ 50 criteria | 88.5 | 100 | 100 | 91.1
  ACR ≥ 70 criteria | 88.5 | 100 | 100 | 86.7
  ACR ≥ 90 criteria | 88.5 | 66.7 | 50 | 76.7
  ACR 100 criteria | 65.4 | 66.7 | 0 | 67.8

6. Primary Outcome: Percentage of Participants Previously Treated With Other Biologics Who Achieved Minimum Response of American College of Rheumatology (ACR) Pediatric 30/50/70/90/100 at Last Assessment of Study
Description: as for outcome 5
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was done in FAS population. Here 'Number of participants analyzed' signifies number of participants with an ACR assessment at the given visit. For arm 'ACZ885 treatment naive: Group 2' there were no participants who had discontinued other biologics due to safety/tolerability issues.
Measure: Number; unit: Percentage of participants
Groups:
- ACZ885 Treatment Naive: Group 1: Participants who were canakinumab treatment- naive and who discontinued other biologics due to lack of efficacy, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treatment Naive: Group 2: Participants who were canakinumab treatment naive and who discontinued other biologics for safety/tolerability reasons, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treatment Naive: Group 3: Participants who were canakinumab treatment naive and who discontinued other biologics for other reasons, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treatment Naive: Group 4: Participants who were canakinumab treatment naive and who never exposed to other biologics, received a s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
Arm/Group | ACZ885 Treatment Naive: Group 1 | ACZ885 Treatment Naive: Group 2 | ACZ885 Treatment Naive: Group 3 | ACZ885 Treatment Naive: Group 4
Number analyzed (Participants) | 30 | 0 | 2 | 89
Percentage of participants
  ACR ≥30 criteria | 96.7 |  | 100 | 91.0
  ACR ≥ 50 criteria | 93.3 |  | 50 | 91.0
  ACR ≥ 70 criteria | 86.7 |  | 50 | 88.8
  ACR ≥ 90 criteria | 83.3 |  | 50 | 77.5
  ACR 100 criteria | 60 |  | 50 | 68.5

7. Secondary Outcome: Percentage of Non--Responders Who Achieved Minimum Response of American College of Rheumatology (ACR) Pediatric 30/50/70/90/100
Description: Adapted ACR Paediatric 30/50/70/90 or 100 was assessed based on following 7 variables: 1.Physician's Global Assessment on a 0-100 mm VAS; 2. Participants Global Assessment on a 0-100 mm VAS; 3. Functional ability; 4. Joints count with active arthritis; 5. Joints count with limitation of motion; 6. Laboratory measure of -CRP and 7. Absence of intermittent fever due to SJIA during the preceding week. Response was defined as ≥ 30%/50%/70%/90% or 100% improvement in at least 3 of the response variables 1 to 6, no intermittent fever (i.e. body temperature ≤ 38°C) in the preceding week (variable 7) and with no more than one variable 1 to 6, worsening by more than 30%.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was done in FAS population. Here 'Number of participants analysed' signifies number of participants with an ACR assessment at the given visit. For arm 'ACZ885 treated: Group 2 (Completed core study)' there were no Non-Responders participants available.
Measure: Number; unit: Percentage of participants
Groups:
- ACZ885 Treated: Group 1 (Discontinued From Core Study): Participants who discontinued from CACZ885G2301 study Part II (NCT00889863), received a subcutaneous (s.c.) injection of canakinumab 4 mg/kg every 4 weeks unless discontinuation occurs. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treated: Group 2 (Completed Core Study): Participants who completed study CACZ885G2301 - Part II (NCT00889863), received an s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
- ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study): Participants who failed to taper their steroid dose in CACZ885G2301 Study -Part I (NCT00889863); received an s.c. injection of canakinumab 4 mg/kg every 4 weeks. Canakinumab 2 mg/kg was administered for participants who were able to taper their steroid dose.
Arm/Group | ACZ885 Treated: Group 1 (Discontinued From Core Study) | ACZ885 Treated: Group 2 (Completed Core Study) | ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study) | ACZ885 Treated: Group 4 (Other Criteria) | ACZ885 Treatment Naive
Number analyzed (Participants) | 17 | 0 | 17 | 6 | 121
Percentage of participants
  ACR ≥30 criteria | 82.4 |  | 76.5 | 83.3 | 92.6
  ACR ≥ 50 criteria | 82.4 |  | 70.6 | 83.3 | 90.9
  ACR ≥ 70 criteria | 82.4 |  | 52.9 | 83.3 | 87.6
  ACR ≥ 90 criteria | 76.5 |  | 23.5 | 50 | 78.5
  ACR 100 criteria | 58.8 |  | 17.6 | 50 | 66.1

8. Secondary Outcome: Percentage of Participants With Minimum Adapted ACR Pediatric ≥ 30 at Baseline Who Achieved Minimum Response of ACR Pediatric 30/50/70/90/100 at Last Assessment of Study
Description: Adapted ACR Paediatric 30/50/70/90 or 100 was assessed based on following 7 variables: 1.Physician's Global Assessment on a 0-100 mm VAS; 2. Participants Global Assessment on a 0-100 mm VAS; 3. Functional ability; 4. Joints count with active arthritis; 5. Joints count with limitation of motion; 6. Laboratory measure of CRP and 7. Absence of intermittent fever due to SJIA during the preceding week. Response was defined as ≥ 30%/50%/70%/90% or 100% improvement in at least 3 of the response variables 1 to 6, no intermittent fever in the preceding week (variable 7) and with no more than one variable 1 to 6 worsening by more than 30%. For minimum adapted ACR paediatric scores, the last measurement recorded from the participant's previous study was considered baseline for the current study.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was done in FAS population. Here 'Number of participants analysed' signifies number of participants with an ACR assessment at the given visit.
Measure: Number; unit: Percentage of participants
Arm/Group | ACZ885 Treated: Group 1 (Discontinued From Core Study) | ACZ885 Treated: Group 2 (Completed Core Study) | ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study) | ACZ885 Treated: Group 4 (Other Criteria)
Number analyzed (Participants) | 16 | 63 | 23 | 5
Percentage of participants
  ACR ≥ 30 | 100 | 100 | 91.3 | 100
  ACR ≥ 50 | 100 | 100 | 87 | 100
  ACR ≥ 70 | 100 | 100 | 78.3 | 100
  ACR ≥ 90 | 100 | 100 | 69.6 | 100
  ACR ≥ 100 | 87.5 | 93.7 | 39.1 | 80

9. Secondary Outcome: Percentage of Participants Able to Taper Oral Steroid Use or Reached Steroid Free Regimen
Description: Steroid tapering with oral steroids was allowed if the participant achieved an adapted ACR Paediatric 50 response and had no fever. A participant was considered to have tapered steroids successfully, if the steroid dose was reduced from baseline and the participant did not flare and maintained a minimum adapted ACR Paediatric 30 at the last measurement. A participant was considered to have unsuccessfully tapered steroids if the steroid dose was reduced during the study but dose at last assessment was equal to or greater than dose at baseline or; if steroid dose was reduced but the participant did not maintain a minimum adapted ACR Paediatric 30 at the last measurement.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was done in FAS population. Here 'Number of participants analysed' signifies number of participants who were steroid users at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | ACZ885 Treated: Group 1 (Discontinued From Core Study) | ACZ885 Treated: Group 2 (Completed Core Study) | ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study) | ACZ885 Treated: Group 4 (Other Criteria) | ACZ885 Treatment Naive
Number analyzed (Participants) | 11 | 9 | 38 | 8 | 71
Percentage of participants
  Steroid free | 36.4 | 55.6 | 23.7 | 25 | 33.8
  Successfully tapered | 27.3 | 0 | 21.1 | 25 | 23.9
  Unsuccessfully tapered | 18.2 | 22.2 | 18.4 | 25 | 11.3
  Did not taper | 18.2 | 22.2 | 36.8 | 25 | 31

10. Secondary Outcome: Number of Participants Who Reduced Their Canakinumab Dose to 2 mg/kg
Description: The canakinumab dose could be reduced from 4 mg/kg to 2 mg/kg in participants who were steroid-free, if requested by the treating physician and agreed by the sponsor. For treatment naive participants , dose reduction was allowed after the participant had received 6 months treatment with canakinumab.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was done in FAS population.
Measure: Number; unit: participants
Arm/Group | ACZ885 Treated: Group 1 (Discontinued From Core Study) | ACZ885 Treated: Group 2 (Completed Core Study) | ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study) | ACZ885 Treated: Group 4 (Other Criteria) | ACZ885 Treatment Naive
Number analyzed (Participants) | 33 | 63 | 40 | 11 | 123
participants | 9 | 29 | 4 | 2 | 18

11. Secondary Outcome: Percentage of Participants With Clinical Remission
Description: Clinical remission was defined as at least 6 months of inactive disease or at least 12 months of inactive disease on medication during the extension period. Participants with inactive disease for at least 6 months, but had loss of inactive disease before 12 months were also determined.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was done in FAS population. Here 'Number of participants analysed' signifies number of participants with an assessment in the given visit.
Measure: Number; unit: Percentage of participants
Arm/Group | ACZ885 Treatment Naive | ACZ885 Treated
Number analyzed (Participants) | 123 | 147
Percentage of participants
  At least 6 consecutive months of inactive disease | 42.3 | 52.4
  At least 12 consecutive months of inactive disease | 26.8 | 42.9
  Loss of inactive disease after 6 months | 8.9 | 6.8

12. Secondary Outcome: Change From Baseline in Disability, Overall Well-Being and Pain Intensity Scores Based on Child Health Assessment Questionnaire (CHAQ) to Last Assessment of Study
Description: The CHAQ was used to assess physical ability, overall well- being and pain intensity experienced by participants. The CHAQ (disability and well-being) dimension consisted of 20 multiple choice items concerning difficulty in performing eight common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and other "activities". Participants were graded for the response in four categories, ranging from 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty) and 3 (unable to do). Participant's pain intensity was assessed by parents and adult participants (18-20 years old) on a VAS scale of 0-100 mm (0 mm: no pain to 100: very severe pain). Change from baseline was calculated by using the formula = (post baseline value - baseline value). For both scales, lower scores indicate increased functional ability.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was performed in FAS population.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | ACZ885 Treated: Group 1 (Discontinued From Core Study) | ACZ885 Treated: Group 2 (Completed Core Study) | ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study) | ACZ885 Treated: Group 4 (Other Criteria) | ACZ885 Treatment Naive
Number analyzed (Participants) | 33 | 63 | 40 | 11 | 121
units on a scale
  Disability score | -0.375 [-2 to 0.625] | 0 [-1.5 to 2.125] | -0.125 [-1.25 to 2.25] | 0 [-2.125 to 1.375] | -0.7143 [-3 to 2.5]
  Overall well-being score | -18 [-64 to 54] | 0 [-36 to 81] | 0 [-36 to 1] | -10 [-69 to 20] | -28 [-100 to 83]
  Pain Intensity score | -13 [-69 to 39] | 0 [-39 to 80] | 0 [-58 to 93] | 0 [-57 to 53] | -39 [-100 to 89]

13. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) Over Time Based on Child Health Questionnaire- Parent Form (CHQ-PF50) to Last Assessment of Study
Description: The Child Health Questionnaire - Parent Form (CHQ-PF50) instrument was used to measure HRQoL aged 5 to 18 years from a parent's perspective. This 14 concept questionnaire measured physical and psychosocial health of the participants on following points: physical functioning, role/social emotional, role/social behavior, role/social physical, bodily pain, general behavior, mental health, self-esteem, general health perception, change in health, parental impact - emotional, parental impact - time, family activities, and family cohesion. Total score ranged from 1-100. Increase in score represented improvement in overall well being of participants. Change from baseline was calculated by using the formula = (post baseline value - baseline value).
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was performed in FAS population. Here 'Number of participants analysed' signifies number of participants with HRQoL assessment in the given visit.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | ACZ885 Treated: Group 1 (Discontinued From Core Study) | ACZ885 Treated: Group 2 (Completed Core Study) | ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study) | ACZ885 Treated: Group 4 (Other Criteria) | ACZ885 Treatment Naive
Number analyzed (Participants) | 26 | 44 | 29 | 8 | 90
units on a scale
  CHQ-PF50 physical score | 14.0407 [-18.289 to 38.33] | 0.6959 [-14.663 to 23.833] | 1.3716 [-42.009 to 41.275] | 13.9255 [-3.074 to 37.083] | 18.8758 [-38.587 to 60.661]
  CHQ-PF50 psychosocial score | 3.8815 [-22.516 to 22.471] | 1.4004 [-14.99 to 30.982] | 0.7582 [-21.674 to 22.907] | 11.9798 [-5.931 to 33.497] | 9.3209 [-23.862 to 48.657]

14. Secondary Outcome: Change From Baseline in EuroQual 5 -Dimension Health Status Questionnaire (EQ-5D) Utility Index and Health State Assessment Scores [EQ Visual Analog Scale (EQ-VAS)] to Last Assessment of Study
Description: EQ-5D HRQoL tool was used for participants above 12 years and EQ-5D proxy for 8-11 years. EQ-5D index scores range from -0.11 (worst possible health, worse than dead), to 0 (dead) to 1 (perfect health). Utility based EQ-5D questionnaire provides generic measure of health for clinical and economic appraisal based on 2 parts: EQ-5D descriptive system - 5 dimensions each with 3 levels (1:no, 2:moderate, 3:severe problem) on: mobility (1=0, 2=0.069, 3=0.314), self-care (1=0, 2=0.104, 3=0.214), usual activities (1=0, 2=0.036, 3=0.094), pain/discomfort (1=0, 2=0, 3=0.386) and anxiety/depression (1=0, 2=0.071, 3=0.2). EQ-5D Total score= 1-0.081-(score of level 2 in present)-0.269 (if at least one of level 3 presents). EQ-5D total score: 1=high quality of life; -0.59 worst quality of life; and EQ-VAS - record participant's self-rated health on vertical, visual analog scale as '100=Best and 0=Worst imaginable health state'.
  Positive change from baseline score indicated improved health status.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was performed in FAS population. Here 'Number of participants analyzed' signifies number of participants with EQ-5D assessment in the given visit.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | ACZ885 Treated: Group 1 (Discontinued From Core Study) | ACZ885 Treated: Group 2 (Completed Core Study) | ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study) | ACZ885 Treated: Group 4 (Other Criteria) | ACZ885 Treatment Naive
Number analyzed (Participants) | 17 | 35 | 22 | 4 | 65
units on a scale
  EQ- 5D Utility Index | 0.204 [-0.636 to 0.945] | 0 [-0.434 to 0.377] | 0.069 [-1.181 to 0.508] | 0.2385 [0 to 0.741] | 0.228 [-0.434 to 1.291]
  EQ-VAS | 21 [-45 to 63] | 0 [-17 to 49] | 5 [-86 to 50] | 28 [0 to 65] | 30 [-24 to 95]

15. Secondary Outcome: Change From Baseline in Pediatric Daytime Sleepiness Scale (PDSS) Score to Last Assessment of Study
Description: Sleep patterns in children and adolescents aged between 11 and 15 years were determined using PDSS instrument to evaluate whether canakinumab helps in reducing sleepiness in children with SJIA. Participants were assessed on 8 items of PDSS, on a scale of 0 to 4 (0 - never, 1 - seldom, 2- sometimes, 3 - frequently and 4 - always). The sum of all the items was reported as total score with a range of 0-32. Change from baseline was calculated by using the formula = (post baseline value - baseline value). A positive change from baseline score indicated improvement.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was performed in FAS population. Here, 'Number of participants analysed' signifies those participants with a value at both baseline and the respective post baseline time point and with an assessment of PDSS score in the given visit..
Measure: Median (Full Range); unit: units on a scale
Arm/Group | ACZ885 Treated: Group 1 (Discontinued From Core Study) | ACZ885 Treated: Group 2 (Completed Core Study) | ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study) | ACZ885 Treated: Group 4 (Other Criteria)
Number analyzed (Participants) | 9 | 12 | 5 | 2
units on a scale | 1 [-9 to 4] | 0.5 [-6 to 9] | 0 [-4 to 6] | -4.5 [-11 to 2]

16. Secondary Outcome: Change From Baseline in Growth Velocity Parameter for Height to Last Assessment of Study
Description: Growth velocity parameter height percentile was determined. Percentile was based on the growth charts smoothed percentile curve released by Centers for Disease control and prevention (CDC) in 2000, by sex and age.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was performed in FAS population. Here, 'Number of participants analyzed' signifies those participants with a value at both baseline and the respective post baseline time point.
Measure: Median (Full Range); unit: Percentile
Arm/Group | ACZ885 Treatment Naive | ACZ885 Treated
Number analyzed (Participants) | 123 | 139
Percentile | -0.01 [-66.18 to 47.06] | 0 [-37.94 to 37.12]

17. Secondary Outcome: Percentage of Participants With Inactive Disease
Description: Inactive disease was defined as no joints with active arthritis; no fever (body temperature ≤ 38 degree Celsius); no rheumatoid rash, serositis, splenomegaly, hepatomegaly, or generalized lymphadenopathy attributable to SJIA; normal CRP, and a rating of no disease activity on the Physician's Global Assessment of disease activity (with a best possible score ≤10 mm on the VAS).
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: The analysis was performed in FAS population. Here 'Number of participants analysed' signifies number of participants with an assessment in the given visit.
Measure: Number; unit: Percentage of participants
Arm/Group | ACZ885 Treated: Group 1 (Discontinued From Core Study) | ACZ885 Treated: Group 2 (Completed Core Study) | ACZ885 Treated: Group 3 (Steroid Taper Failures in Core Study) | ACZ885 Treated: Group 4 (Other Criteria) | ACZ885 Treatment Naive
Number analyzed (Participants) | 33 | 63 | 40 | 11 | 122
Percentage of participants | 39.4 | 79.4 | 12.5 | 36.4 | 50.8

18. Secondary Outcome: Change From Baseline in Growth Velocity Parameters to Last Assessment of Study
Description: Growth velocity parameter weight percentile was determined. Percentile was based on the growth charts smoothed percentile curve released by Centers for Disease control and prevention (CDC) in 2000, by sex and age.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: as for outcome 16
Measure: Median (Full Range); unit: Percentile
Arm/Group | ACZ885 Treatment Naive | ACZ885 Treated
Number analyzed (Participants) | 123 | 139
Percentile | 0.1 [-47.35 to 82.84] | 0 [-62.49 to 56.87]

19. Secondary Outcome: Change From Baseline in Growth Velocity Parameter for BMI to Last Assessment of Study
Description: Growth velocity parameter BMI percentile was determined. Percentile was based on the growth charts smoothed percentile curve released by Centers for Disease control and prevention (CDC) in 2000, by sex and age.
Time Frame: Baseline up to last assessment (4 years) or date of discontinuation, which ever occurred earlier
Population: as for outcome 16
Measure: Median (Full Range); unit: Percentile
Arm/Group | ACZ885 Treatment Naive | ACZ885 Treated
Number analyzed (Participants) | 123 | 139
Percentile | 1.08 [-66.95 to 76.3] | -0.77 [-72.88 to 88.47]

ADVERSE EVENTS:
Time Frame: From start of study treatment (Day 1) to end of follow-up period (Week 271)
Description: The analysis was performed in safety set, defined as all subjects who received at least one dose of study drug under this study protocol.
Arm/Group | ACZ885 Treated | ACZ885 Treatment Naive
Serious Adverse Events (participants affected / at risk) | 47/147 | 40/123
Other Adverse Events (participants affected / at risk) | 124/147 | 91/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 Treated (N=147) | ACZ885 Treatment Naive (N=123)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 10 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Device dislocation (General disorders) | 0 | 1
Disease progression (General disorders) | 1 | 0
Drug ineffective (General disorders) | 1 | 1
Injury associated with device (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 4
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abscess neck (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 4 | 2
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Gastroenteritis yersinia (Infections and infestations) | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Impetigo (Infections and infestations) | 1 | 0
Infected bites (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lymph node abscess (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1
Parvovirus infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 3
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pseudocroup (Infections and infestations) | 1 | 0
Salmonella sepsis (Infections and infestations) | 0 | 1
Scarlet fever (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 2 | 0
Tonsillitis streptococcal (Infections and infestations) | 2 | 0
Toxoplasmosis (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 3 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 1
Liver function test abnormal (Investigations) | 1 | 0
Serum ferritin increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 14 | 13
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Superior sagittal sinus thrombosis (Nervous system disorders) | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 2
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 Treated (N=147) | ACZ885 Treatment Naive (N=123)
Ear pain (Ear and labyrinth disorders) | 10 | 7
Abdominal pain (Gastrointestinal disorders) | 21 | 22
Abdominal pain upper (Gastrointestinal disorders) | 18 | 13
Diarrhoea (Gastrointestinal disorders) | 30 | 16
Nausea (Gastrointestinal disorders) | 17 | 11
Vomiting (Gastrointestinal disorders) | 35 | 18
Fatigue (General disorders) | 10 | 3
Pyrexia (General disorders) | 38 | 27
Bronchitis (Infections and infestations) | 13 | 6
Conjunctivitis (Infections and infestations) | 8 | 6
Gastroenteritis (Infections and infestations) | 28 | 19
Influenza (Infections and infestations) | 14 | 4
Nasopharyngitis (Infections and infestations) | 47 | 32
Oral herpes (Infections and infestations) | 11 | 1
Otitis media (Infections and infestations) | 11 | 7
Pharyngitis (Infections and infestations) | 15 | 15
Respiratory tract infection (Infections and infestations) | 7 | 13
Rhinitis (Infections and infestations) | 35 | 26
Tonsillitis (Infections and infestations) | 10 | 7
Upper respiratory tract infection (Infections and infestations) | 36 | 24
Urinary tract infection (Infections and infestations) | 8 | 4
Viral infection (Infections and infestations) | 6 | 11
Viral upper respiratory tract infection (Infections and infestations) | 10 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 9 | 12
Contusion (Injury, poisoning and procedural complications) | 11 | 0
Fall (Injury, poisoning and procedural complications) | 11 | 7
Ligament sprain (Injury, poisoning and procedural complications) | 11 | 5
Alanine aminotransferase increased (Investigations) | 8 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 25
Arthritis (Musculoskeletal and connective tissue disorders) | 9 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 9
Joint swelling (Musculoskeletal and connective tissue disorders) | 9 | 5
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 23 | 27
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 12
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 4
Headache (Nervous system disorders) | 30 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 28
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 36 | 17
Eczema (Skin and subcutaneous tissue disorders) | 12 | 16
Rash (Skin and subcutaneous tissue disorders) | 15 | 13
Urticaria (Skin and subcutaneous tissue disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (i.e, data from all sites) in the clinical trial.